CLINICAL TRIAL: NCT00283075
Title: Use of Mouse Renal Adenocarcinoma Cell-containing Agarose-agarose Macrobeads in the Treatment of Patients With End-stage, Treatment-resistant Epithelial-derived Cancer
Brief Title: Mouse Cancer Cell-containing Macrobeads in the Treatment of Human Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0407007343
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Intraabdominal Cancers (Various Types)
Keywords: intraabdominal cancer (carcinomas); agarose macrobeads; mouse kidney cancer cells; cancer cell growth inhibition
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cancer macrobeads (Experimental): Cancer Macrobead placement in abdominal cavity
  Interventions: Biological: Cancer Macrobead placement in abdominal cavity

INTERVENTIONS:
Biological: Cancer Macrobead placement in abdominal cavity — 8 macrobeads per kg
  Other Names: cancer macrobead

SUMMARY:
This is a phase 1 trial to evaluate the safety and toxicity of mouse kidney cancer cell-containing agarose-agarose macrobeads that are implanted in the abdominal cavity as a proposed biological treatment of patients with end-stage, treatment-resistant cancer. The macrobeads have been extensively tested in tumor models in mice and rats, as well as in forty-five veterinary patients (cats and dogs) with naturally occurring tumors of various types including breast cancer, prostate cancer, liver cancer, and lymphoma with clear tumor responses and no significant detectable toxicity.

DETAILED DESCRIPTION:
Cancer in its various forms continues to be a major U.S. health problem, accounting for 550,000 deaths a year, as well as much disability and suffering. Treatment for cancer has traditionally consisted of three modalities: surgery, radiation therapy, and chemotherapy. Advances with all three modalities over the years have produced long-term remissions and/or cures in certain types of cancer such as the leukemias, and prolonged survival for many other patients. Much remains to be accomplished, however, especially with respect to the treatment of solid tumors, including some of the most common cancers such as those of the lung, colon, breast, ovary, prostate and kidney. New types of less toxic and debilitating therapy are needed.

Among the therapeutic possibilities currently being explored, those that involve biological control mechanisms seem both promising and attractive. Although it has long been thought that cancer cells are not subject to the same regulatory growth control mechanisms that function in normal cells, there is a substantial body of evidence that they can respond to feedback signals telling them to slow or stop their growth. In addition, it has been determined that a relatively small population of cells within a tumor (cancer "stem" or progenitor cells) are responsible for continued tumor growth and that it is these cells that must be controlled if biological anti-tumor therapy is to be effective.

The proposed cancer treatment being tested in this Phase 1 clinical trial is based on the concept that tumor growth can be controlled by tumor mass or signals that indicate that such mass is present. In this case, however, the induction of the growth-slowing signals is brought about not by tumor mass, but by placing mouse kidney cancer cells in an agarose matrix, which both selects for cancer progenitor cells and also causes them to produce and release signals that inhibit the growth of freely growing cancer cells of the same or different type in a laboratory dish or in a tumor-bearing animal or human (i.e. is also not species-specific). This approach has proven both safe and effective in animal models and veterinary patients, and it is now in the first stage of human testing. With Phase 1 completed, we are now implementing Phase 2 efficacy trials that for the present are focused on colorectal cancer, pancreatic cancer, and prostate cancer. The Phase 1 trial remains open to a range of epithelial-derived cancer.

ELIGIBILITY:
Inclusion Criteria:

* End-stage, treatment resistant epithelial-derived cancer (carcinoma) arising originally within the abdominal cavity with expected minimum six-month survival

Exclusion Criteria:

* Multiple intraabdominal metastases or carcinomatosis or other medical conditions indicating that the procedure would be of too high a risk for the individual

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-01; Primary Completion 2012-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry H Smith, MD, PhD, Principal Investigator — The Rogosin Institute
Locations (1):
- NewYork Presbyterian Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeWys WD. Studies correlating the growth rate of a tumor and its metastases and providing evidence for tumor-related systemic growth-retarding factors. Cancer Res. 1972 Feb;32(2):374-9. No abstract available. PMID 4258017
- [Background] Fisher B, Gunduz N, Coyle J, Rudock C, Saffer E. Presence of a growth-stimulating factor in serum following primary tumor removal in mice. Cancer Res. 1989 Apr 15;49(8):1996-2001. PMID 2702641
- [Background] Prehn RT. The inhibition of tumor growth by tumor mass. Cancer Res. 1991 Jan 1;51(1):2-4. PMID 1988084
- [Background] Reya T, Morrison SJ, Clarke MF, Weissman IL. Stem cells, cancer, and cancer stem cells. Nature. 2001 Nov 1;414(6859):105-11. doi: 10.1038/35102167. PMID 11689955
- [Background] Al-Hajj M, Wicha MS, Benito-Hernandez A, Morrison SJ, Clarke MF. Prospective identification of tumorigenic breast cancer cells. Proc Natl Acad Sci U S A. 2003 Apr 1;100(7):3983-8. doi: 10.1073/pnas.0530291100. Epub 2003 Mar 10. PMID 12629218
- [Background] Smith BH, Gazda LS, Conn BL, Jain K, Asina S, Levine DM, Parker TS, Laramore MA, Martis PC, Vinerean HV, David EM, Qiu S, North AJ, Couto CG, Post GS, Waters DJ, Cordon-Cardo C, Hall RD, Gordon BR, Diehl CH, Stenzel KH, Rubin AL. Hydrophilic agarose macrobead cultures select for outgrowth of carcinoma cell populations that can restrict tumor growth. Cancer Res. 2011 Feb 1;71(3):725-35. doi: 10.1158/0008-5472.CAN-10-2258. Epub 2011 Jan 24. PMID 21266362
- [Background] Smith BH, Gazda LS, Conn BL, Jain K, Asina S, Levine DM, Parker TS, Laramore MA, Martis PC, Vinerean HV, David EM, Qiu S, Cordon-Cardo C, Hall RD, Gordon BR, Diehl CH, Stenzel KH, Rubin AL. Three-dimensional culture of mouse renal carcinoma cells in agarose macrobeads selects for a subpopulation of cells with cancer stem cell or cancer progenitor properties. Cancer Res. 2011 Feb 1;71(3):716-24. doi: 10.1158/0008-5472.CAN-10-2254. Epub 2011 Jan 24. PMID 21266363
- [Background] Gazda LS, Martis PC, Laramore MA, Bautista MA, Dudley A, Vinerean HV, Smith BH. Treatment of agarose-agarose RENCA macrobeads with docetaxel selects for OCT4(+) cells with tumor-initiating capability. Cancer Biol Ther. 2013 Dec;14(12):1147-57. doi: 10.4161/cbt.26455. Epub 2013 Sep 12. PMID 24025409

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-six subjects provided informed consent to participate in this study; of these 31 subjects underwent the implantation of macrobeads that contain mouse renal adenocarcinoma cells (RENCA macrobeads). The first subject was implanted on 6 April 2005 and the last subject was implanted on 1 November 2011.
Groups:
- 8 RENCA Macrobeads/kg Body Weight Implantation: RENCA macrobeads placement in abdominal cavity at 8 RENCA macrobeads/kg body weight.
- 16 RENCA Macrobeads/kg Body Weight Implantation: RENCA macrobeads placement in abdominal cavity at 16 RENCA macrobeads/kg body weight.
Period: Overall Study
Arm/Group | 8 RENCA Macrobeads/kg Body Weight Implantation | 16 RENCA Macrobeads/kg Body Weight Implantation
Started | 25 | 6
Completed | 25 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who had at least one implantation of RENCA macrobeads, either at 8 RENCA macrobeads/kg body weight or 16 RENCA macrobeads/kg body weight.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 15
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12
  Hispanic | 2
  Asian | 1
  Not Available | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of RENCA Macrobeads
Description: Dose limiting toxicity (DLT) was defined as:
  * any Grade 2 allergic reaction of generalized urticaria or any other Grade ≥ 3 allergic reaction;
  * any Grade ≥ 3 infection and
  * any Grade ≥ 3 local (intraperitoneal) reaction and any Grade ≥ 3 hematologic or non- hematologic reaction.
  This definition of DLT is in accord with the NCI CTCAE v3.0.
  Maximum tolerated dose (MTD) was to be identified if, within a cohort, > 1 subject out of the first 3, or 2 subjects out of 5 experienced DLT. In such a case, the MTD will have been exceeded, and the administration of the study agent was to cease. MTD would not be considered to have been reached if no DLTs were observed.
Time Frame: 6 months
Measure: Number; unit: RENCA Macrobeads/kg
Arm/Group | All Participants
Number analyzed (Participants) | 31
RENCA Macrobeads/kg | NA — MTD of of RENCA macrobeads has not been reached because no DLTs were observed.

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was measured as date of first implantation to date of death of any cause, and was analyzed using the Kaplan-Meier method.
Time Frame: From date of RENCA macrobeads implantation until date of death from any cause
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Participants: All participants who had at least one implantation of RENCA macrobeads, either at 8 macrobeads/kg body weight or 16 macrobeads/kg body weight.
Arm/Group | All Participants
Number analyzed (Participants) | 31
months
  All Cancer Type | 5.4 [2.2 to 7.0]
  Colorectal Cancer | 7.0 [1.1 to 9.7]
  Pancreatic Cancer | 1.1 [1.0 to 2.2]
  Other Cancer | 5.7 [2.0 to 7.0]

3. Other Pre Specified Outcome: Tumor Marker Response
Description: Tumor marker response after the first implantation with RENCA macrobeads. Responders showed at least a 20% decrease from baseline in Cancer Antigen 19-9 (CA19-9) or Carcinoembryonic Antigen (CEA); Non-responders do not show at least a 20% decrease from baseline in CA19-9 or CEA.
Time Frame: Prior to Implantation and Day 7, Day 14, Day 21 and Day 28 after each implantation
Population: All participants who had at least one implantation of RENCA macrobeads, either at 8 macrobeads/kg body weight or 16 macrobeads/kg body weight.
Measure: Number; unit: participants
Groups:
- Day 7: Tumor marker response at Day 7 after the first implantation.
- Day 14: Tumor marker response at Day 14 after the first implantation.
- Day 21: Tumor marker response at Day 21 after the first implantation.
- Day 28: Tumor marker response at Day 28 after the first implantation.
Arm/Group | Day 7 | Day 14 | Day 21 | Day 28
Number analyzed (Participants) | 20 | 21 | 13 | 17
participants
  Responder | 5 | 13 | 9 | 10
  Non-Responder | 15 | 8 | 4 | 7

4. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: Dose limiting toxicity (DLT) was defined as:
  * any Grade 2 allergic reaction of generalized urticaria or any other Grade ≥ 3 allergic reaction;
  * any Grade ≥ 3 infection and
  * any Grade ≥ 3 local (intraperitoneal) reaction and any Grade ≥ 3 hematologic or non- hematologic reaction.
  This definition of DLT is in accord with the NCI CTCAE v3.0.
Time Frame: 6 months
Measure: Number; unit: Participants who observed DLT
Arm/Group | 8 RENCA Macrobeads/kg Body Weight Implantation | 16 RENCA Macrobeads/kg Body Weight Implantation
Number analyzed (Participants) | 25 | 6
Participants who observed DLT | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 20/31
Other Adverse Events (participants affected / at risk) | 27/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=31)
Implant site fluid collection (Surgical and medical procedures) | 1 (1)
Tear from mesh s/p hernia repair (Surgical and medical procedures) | 1 (1)
Intermittent fever (General disorders) | 1 (1)
Disease progression (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hypophagia (General disorders) | 1 (1)
Pleurodesis (General disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hypotension, poor nutrition (General disorders) | 1 (1)
Aspiration (General disorders) | 1 (1)
Jaundice (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Transfusion (General disorders) | 1 (2)
Dehydration (General disorders) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Blood creatinine increased (General disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Melena (Gastrointestinal disorders) | 1 (1)
Hypotension (General disorders) | 1 (1)
Anemia (General disorders) | 1 (1)
Incision site pain (Surgical and medical procedures) | 1 (1)
Wound complication (Surgical and medical procedures) | 1 (1)
Hyponatremia (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Hydronephrosis (General disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=31)
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 2
Fatigue (General disorders) | 15
Inflammation (General disorders) | 4
Pain (General disorders) | 5
Pyrexia (General disorders) | 11
Incision site pain (Injury, poisoning and procedural complications) | 3
Hemoglobin decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Night sweats (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 4
Umbilical erythema (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes